CLINICAL TRIAL: NCT05472311
Title: Implementation and Scale Up of a Single-visit, Screen-and-treat Approach With Thermal Ablation for Sustainable Cervical Cancer Prevention Services in Kenya
Brief Title: Cervical Cancer Elimination -Using Implementation Science to Evaluate Deliver and Cost Introduction of Thermal Ablation
Acronym: TIBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Nelly Mugo, Research Associate Professor: Global Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014200; R01CA258590-01 (NIH)
Record Dates: First submitted 2022-06-10; First posted 2022-07-25 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cervical Cancer
Keywords: invasive cervical cancer; cervical intra-epithelial lesion (CIN); human papillomavirus; single visit screen- and - treat (SVA-SAT); thermal ablation; implementation science
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: Using implementation science methods to evaluate the implementation of thermal ablation for treatment of pre-cancer lesions of the cervix in reproductive health clinics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treat with thermal ablation (Other): Women who screen positive for pre-cancer lesions of the cervix will be offered treatment with thermal ablation and the process of implementation evaluated using implementation science RE-AIM framework
  Interventions: Other: Thermal Ablation

INTERVENTIONS:
Other: Thermal Ablation — Thermal ablation is based on local heating (around 100 degrees centigrade), applied for 20 to 60 seconds to destroy abnormal tissue by burning and inducing necrosis of pre-cancer and surrounding tissue. It has been used in by gynecological surgery for over 50 years, proven safe and easy to use by middle level health care providers in primary care settings.
  Other Names: TA

SUMMARY:
Global elimination of cervical cancer is a feasible goal; however, the countries with the greatest disease burden also have the greatest healthcare system challenges. Cervical cancer (CC) is almost entirely preventable, yet, it remains the 2nd most common cause of cancer and is the most common cause of cancer deaths among women in the majority of Low-Middle-Income-Countries (LMIC) including Kenya. Effective low-cost interventions for early detection of pre-cancer lesions have been available but there remains very low coverage with about 16% eligible women screened in Kenya. Cryotherapy has been introduced as a low-cost intervention for treatment of pre-cancer lesions, however, challenges with equipment shortage, costs, supply chain difficulties of refrigerant gas and equipment failure health facilities has been cited as a reason for the low treatment rates of screen positive women. In Kenya only about 30% of women screening positive access treatment for the pre-cancer lesions. This project will introduce thermal ablation (TA), which is proven to be safe and as effective as cryotherapy for treatment of pre-cancer lesions of the cervix. TA uses electricity, batteries or solar to charge, takes a shorter time to use, is a small easily portable equipment.

The primary aim of the study is to deliver, evaluate and cost implementation of the 'Single Visit Screen and Treat with Thermal Ablation' (SVA-SAT+TA) intervention for treatment of women who screen positive for pre-cancer lesions of the cervix in reproductive health clinics in Kenya, using implementation science framework to inform National scale-up.

To achieve national and global goals to eliminate cervical cancer, there is an urgent need to adapt, implement, and scale-up effective technologies in Kenya. The proposed research project will develop a contextually appropriate implementation and dissemination model to guide effective scale-up of the single visit screen and treat approach with use of thermal ablation to health facilities to bridge access to cervical cancer prevention services for women in Kenya and similar low resource settings.

DETAILED DESCRIPTION:
The mainstay of cervical cancer (CC) prevention in low- and middle-income counties (LMIC) has been the single-visit approach with screen-and-treat (SVA-SAT) method, using visual inspection with acetic acid (VIA) and ablative treatment with cryotherapy to manage precancerous lesions. It is a low-cost screening approach and minimizes loss to follow-up compared to traditional cytology. In Kenya, there is extremely low fidelity of SVA-SAT. Thermal ablation (TA) is an effective alternative to cryotherapy for ablation of precancerous lesions, and has been recommended by the World Health Organization (WHO) since 2019. Preliminary data from an investigative team member demonstrated safety, effectiveness, and acceptability to women when delivered by nurses in Zambia and Kenya. The portable device can be charged with electricity, batteries or solar panels, which is ideal for low-resource settings. Successful implementation and scale-up of TA within the SVA-SAT approach could optimize CC prevention.

This is a five-year prospective, stepped-wedge, cluster randomized trial to implement SVA-SAT+TA in 10 reproductive health (RH) clinics in central Kenya. The study uses mixed-methods evaluation based on the RE-AIM (Reach, Effectiveness, Adoption, Implementation and Maintenance) framework to assess the intervention's impact.

In collaboration with multi-level (clinic, county, national) stakeholders this project will develop a sustainable D&I strategy and leverage trial implementation to include costing and budget impact analysis. The objective is to develop and evaluate a locally contextualized dissemination and implementation (D&I) strategy for SVA-SAT with TA (SVA-SAT+TA) to inform national scale-up. The hypothesis is that TA will enhance the feasibility, adoption, and sustainability of CC prevention services via SVA-SAT, compared to the standard of care with cryotherapy.

Design:

Prospective, stepped-wedge, cluster randomized trial to implement SVA-SAT+TA in ten reproductive health (RH) clinics in central Kenya.

Population: Mixed population: Reproductive health care workers, health manager's, women seeking services for cervical cancer screening and women who screen positive for pre-cancerous lesions of the cervix.

Objective 1:

Develop a dissemination and implementation strategy to introduce SVA-SAT+TA that effectively accounts for the heterogeneity of the client, provider, and system inputs.

Approach: The project will use qualitative interviews with women seeking CC prevention services, reproductive health (RH) providers, RH managers, and key program stakeholders to identify actionable barriers and facilitators to SVA-SAT+TA uptake. These data will be presented at a stakeholder workshop to synthesize and contextualize strategies to effectively introduce the intervention and provide guidance for scale up.

Objective 2:

Deliver the SVA-SAT+TA intervention at scale in RH clinics and evaluate implementation using the RE-AIM framework.

Approach: The SVA-SAT+TA will be introduced into RH clinics using a stepped-wedge study design and using RE-AIM framework the process will be rigorously evaluated on how effective it is disseminated and implemented. Key endpoints will include:

1. (REACH) Proportion of the clinics reached, providers trained;
2. (EFFECTIVENESS) Intervention effect on SVA-SAT process measures: number of screen positive women identified per month, treatment completion rate compared to pre-intervention, and the patient-level TA fidelity of implementation assessed by testing Human Papillomavirus (HPV) clearance
3. (ADOPTION) Proportion of the clinics incorporating TA into routine care
4. (IMPLEMENTATION) Describe drivers of success/failure using the Consolidated Framework for Implementation Research (CFIR)
5. (MAINTENANCE) Proportion of clinics that continue to provide and sustain SVA-SAT+TA services post intervention implementation.

Objective 3:

Compare the cost and budget impact of SVA-SAT+TA to SVA-SAT using cryotherapy. Approach: Using micro-costing techniques to quantify the programmatic costs of SVA-SAT with cryotherapy and with TA.

ELIGIBILITY:
Inclusion Criteria:

* Policy makers
* Health facility managers
* Health care providers at participating reproductive health clinics
* Women seeking cervical cancer screening services
* Women who screen positive for pre-cancer lesion of the cervix
* Consent to study participation
* Age 25-60 years
* Women seeking cervical cancer screening services at participating RH clinics
* Health care providers providing cervical cancer prevention services at participating RH clinics

Exclusion Criteria:

-Any individual who declines to participate or have their data collected for purpose of research

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 565 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Index of barriers to introduction of SAT_SVA+TA | 3 months
  Using a participatory approach through engagement of key stakeholders (women seeking cervical cancer prevention services, frontline health care workers, managers and policy makers) describe factors that deter successful introduction and scalability of SAT-SVA+TA intervention
Index of facilitators to introduction of SAT_SVA+TA | 3 months
  Using a participatory approach through engagement of key stakeholders (women seeking cervical cancer prevention services, frontline health care workers, managers and policy makers) describe factors that make it suitable for successful introduction and scalability of SAT-SVA+TA intervention
Deliver and Using the RE-AIM Framework Evaluate the Implementation of Thermal Number of providers trained who continue to provide treatment for pre-cancer lesions of the cervix using thermal ablation with a single visit approach | 4 years
  The number of providers trained who continue to provide treatment for pre-cancer lesions of the cervix using thermal ablation with a single visit approach during the periods before, during and after introduction of TA to RH clinics
Impact of the SVA-SAT+TA on effective uptake of treatment of pre-cancer lesions of the cervix | 4 years
  Measure treatment completion rate compared to pre-intervention for women who screen positive for pre-cancer lesions of the cervix
Sustained use of TA to treat pre cancer lesions of the cervix in RH clinics in Kenya | 4 years
  The treatment completion rates of women with pre-cancer lesions of the cervix after withdrawal of active implementation support by project personnel
HPV Clearance post treatment with TA | 6 months after treatment
  The number of screen positive women treated with TA that clear HPV infection post treatment

SECONDARY OUTCOMES:
Cost impact of SVA-SAT_TA | 4 years
  Quantify the programmatic costs of SVA-SAT for treatment of pre-cancer lesions of the cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mugo, MPH, MMed, Principal Investigator — University of Washington
Locations (1):
- Phrd-Ccr-Kemri, Thika, Kiambu County, Kenya

IPD SHARING:
Plan to Share IPD: No
De-identified provider interviews will be shared with other Implementation Science researchers to improve healh care outcomes.

REFERENCES:
- [Derived] Adhiambo HF, Thomas K, Coe MM, Oluoch L, Ihaji V, Kerubo MB, Kinyua A, Njoroge S, Ngure K, Shin M, Odeny TA, Weiner B, Mugo N, Gimbel S. Applying FRAME-IS to Characterize Provider-led Adaptations to a Cervical Cancer Prevention Intervention in Kenya. Res Sq [Preprint]. 2025 Jul 15:rs.3.rs-6933921. doi: 10.21203/rs.3.rs-6933921/v1. PMID 40709265
- [Derived] Shin MB, Oluoch LM, Barnabas RV, Baynes C, Fridah H, Heitner J, Kerubo MB, Ngure K, Pinder LF, Thomas KK, Mugo NR, Gimbel S. Implementation and scale-up of a single-visit, screen-and-treat approach with thermal ablation for sustainable cervical cancer prevention services: a protocol for a stepped-wedge cluster randomized trial in Kenya. Implement Sci. 2023 Jun 26;18(1):26. doi: 10.1186/s13012-023-01282-3. PMID 37365575